CLINICAL TRIAL: NCT01697137
Title: Patient and Physician Intervention to Increase Organ Donation in Primary Care Settings
Brief Title: Patient and Physician Intervention to Increase Organ Donation
Acronym: DECIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Daryl Thornton, Assistant Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 6 R39OT22056-01-01; R39OT22056 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Tissue and Organ Donation; Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Following enrollment, participants will visit with their primary care provider per usual.
- Participant Video and Provider Cueing (Experimental): Participants will watch a video prior to meeting with their provider. Participants will then cue their providers to discuss organ donation with them.
  Interventions: Behavioral: Participant Video and Provider Cueing

INTERVENTIONS:
Behavioral: Participant Video and Provider Cueing — Participants will watch a 5-minute video and then select a question about donation to discuss with their primary care provider (provider cueing).
  Arms: Participant Video and Provider Cueing

SUMMARY:
The number of persons on the national solid organ waiting list continues to increase while the number of donated organs has failed to keep pace. In some portions of northeastern Ohio the donation rate is as low as 32%. There is a positive association between discussing organ donation with a primary care physician and signing a donor card. However, such discussions are rare. The investigators propose a blinded randomized controlled trial to evaluate the effectiveness of two interventions: 1) showing a donation video to patients in primary care settings waiting to see their physician and 2) cueing of primary care providers to have donation discussions with their patients. The study will be conducted throughout Cuyahoga County in at least 10 ambulatory clinics associated with a single county medical system. Nine hundred patients over 15.5 years of age will be enrolled. The investigators hypothesize that patients exposed to the interventions will be 1) more likely to consent to donate organs, 2) more likely to have donation discussions with their primary care providers, and 3) equally satisfied with the time spent with their doctor compared to patients who are not exposed to the interventions.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 visits with their primary care provider in the last 3 years
* Not previously consented to organ donation
* At least 15.5 years of age
* Less than 78 years of age

Exclusion Criteria:

* Visually impaired
* Cognitively impaired
* Non-English speaking

Ages: 15 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 916 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who consent to donate organs | 1 Day
  Consent either on the electronic donor registry or by completion of a organ donor card.

SECONDARY OUTCOMES:
Proportion of participants who reported holding donation discussions with their primary care provider | 1 Day

OTHER OUTCOMES:
Proportion of participants who were satisfied with time spent with their provider on the study date | 1 Day
  Proportion of participants who were somewhat or very satisfied with the amount of time spent with their provider during the date of the study.

CONTACTS AND LOCATIONS:
Overall Officials: John D Thornton, MD, MPH, Principal Investigator — Case Western Reserve University
Locations (1):
- The MetroHealth System, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Thornton JD, Sullivan C, Albert JM, Cedeno M, Patrick B, Pencak J, Wong KA, Allen MD, Kimble L, Mekesa H, Bowen G, Sehgal AR. Effects of a Video on Organ Donation Consent Among Primary Care Patients: A Randomized Controlled Trial. J Gen Intern Med. 2016 Aug;31(8):832-9. doi: 10.1007/s11606-016-3630-5. PMID 26921161